CLINICAL TRIAL: NCT00002123
Title: A Double-Blind, Randomized, Comparative Study of Delavirdine Mesylate (U-90152S) in Combination With Didanosine (ddI) Versus ddI Alone in HIV-1 Infected Individuals With CD4 Counts of <= 300/mm3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacia and Upjohn (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 228A; M/3331/0017
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-11

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Delavirdine; Didanosine

INTERVENTIONS:
Drug: Delavirdine mesylate
Drug: Didanosine

SUMMARY:
To evaluate the safety, tolerance, pharmacokinetics, and efficacy of delavirdine mesylate (U-90152S) in combination with didanosine (ddI) versus ddI alone in HIV-positive patients.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* AZT.

Patients must have:

* HIV-1 seropositivity.
* CD4 count <= 300 cells/mm3.
* No active or acute (onset within the past month) opportunistic infections such as active cryptococcosis, pneumocystis carinii, herpes zoster, histoplasmosis, or cytomegalovirus (CMV).
* Consent of parent or guardian if less than 18 years of age.
* Understanding of potential risk to fetus related to study participation.
* Acceptable medical history, physical exam, EKG, and chest x-ray during screening.

NOTE:

* Patients with cutaneous Kaposi's sarcoma requiring no systemic therapy are permitted.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Active tuberculosis that is sensitive to rifampin.
* Inability to swallow numerous tablets.
* Clinically significant active or acute medical problems, including progressive multifocal leukoencephalopathy, lymphoma, or malignancy requiring systemic therapy.
* Clinically significant hypersensitivity to piperazine-type drugs (e.g., Antepar and Stelazine).
* Grade 2 or worse baseline organ function. NOTE:
* Hemophiliacs with grade 2 bilirubin, alkaline phosphatase, SGOT, or SGPT will be considered if these values have been stable over the past year. NOTE:
* Patients with suspected Gilbert's syndrome will be considered if bilirubin is grade 2 or better.

Patients with the following prior conditions are excluded:

* History of pancreatitis within the past 2 years.
* History of clinically significant nervous system or muscle disease, seizure disorder, AIDS dementia, or psychiatric disorder that would preclude study compliance.
* History of grade 2 or worse peripheral neuropathy.
* Intolerance to ddI in previous treated patients.

Prior Medication:

Excluded:

* More than 4 months total of prior ddI.
* Any prior ddC, d4T, or 3TC.
* Prior nonnucleoside reverse transcriptase inhibitors, including L-drugs, nevirapine, TIBO, HEPT, delavirdine, atevirdine, and alpha-APA.
* Other investigational antiretroviral medications (including foscarnet) or immunomodulators (including all interferons) within 21 days prior to initial study drug dose.
* Prior prophylactic or therapeutic HIV-1 gp120 or 160 vaccines.
* Rifampin, rifabutin, astemizole, loratadine, or terfenadine within 21 days prior to initial study drug dose.
* Any unapproved investigational medication for any indication within 21 days prior to initial study drug dose.

Required:

* AZT therapy at some time prior to screening. Active substance abuse.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (84):
- United States (83):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - East Bay AIDS Ctr, Berkeley, California
  - California Med Research Group, Fresno, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Los Angeles County / Health Research Assoc / Drew Med Ctr, Los Angeles, California
  - CARE Ctr / UCLA Med Ctr, Los Angeles, California
  - UCI Med Ctr, Orange, California
  - AIDS Community Research Consortium, Redwood City, California
  - UCD Med Ctr / AIDS and Related Disorders Clinic, Sacramento, California
  - St Lukes Medical Group, San Diego, California
  - UCSD / Ctr for Special Immunology, San Diego, California
  - ViRx Inc, San Francisco, California
  - Saint Francis Mem Hosp, San Francisco, California
  - Davies Med Ctr, San Francisco, California
  - Shared Med Research Foundation, Tarzana, California
  - Harbor - UCLA Med Ctr, Torrance, California
  - Univ Hosp / Univ of Colorado Health Sci Ctr, Denver, Colorado
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - Caremark Inc, Palm Beach Gardens, Florida
  - Infectious Disease Research Institute Inc, Tampa, Florida
  - Infectious Disease Rsch Consortium of GA / SE Clin Resources, Atlanta, Georgia
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Univ of Illinois, Chicago, Illinois
  - Indiana Univ Infectious Disease Research Clinic, Indianapolis, Indiana
  - Univ of Iowa, Iowa City, Iowa
  - Univ of Kansas School of Medicine / Univ Hosp, Kansas City, Kansas
  - Univ of Kansas School of Medicine, Wichita, Kansas
  - Univ of Kentucky Med Ctr / Chandler Med Ctr, Lexington, Kentucky
  - Tulane Univ Med School, New Orleans, Louisiana
  - AIDS Consultation Service / Maine Med Ctr, Portland, Maine
  - Univ of Maryland at Baltimore, Baltimore, Maryland
  - Massachusetts Gen Hosp, Boston, Massachusetts
  - Brigham and Women's Hosp, Boston, Massachusetts
  - Boston City Hosp / FGH-1, Boston, Massachusetts
  - New England Deaconess Hosp, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Univ of Massachusetts Med Ctr, Worcester, Massachusetts
  - Univ of Michigan Hospitals and Health Ctrs, Ann Arbor, Michigan
  - Harper Hosp, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - St Paul Ramsey Med Ctr / HIV Program Office, Saint Paul, Minnesota
  - Univ of Missouri at Kansas City School of Medicine, Kansas City, Missouri
  - Washington Univ, St Louis, Missouri
  - Univ of Nebraska Med Ctr / HIV Clinic, Omaha, Nebraska
  - Jersey Shore Med Ctr, Neptune City, New Jersey
  - Albany Med College, Albany, New York
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Community Research Initiative on AIDS, New York, New York
  - Beth Israel Med Ctr, New York, New York
  - Saint Vincent's Hosp and Med Ctr, New York, New York
  - New York Hosp - Cornell Med Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Community Health Network, Rochester, New York
  - Univ of Rochester Med Ctr, Rochester, New York
  - SUNY / Health Sciences Ctr at Stony Brook, Stony Brook, New York
  - New York Med College / Westchester County Med Ctr, Valhalla, New York
  - Univ of North Carolina School of Medicine, Chapel Hill, North Carolina
  - Carolinas Med Ctr, Charlotte, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Univ of Cincinnati / Holmes Hosp, Cincinnati, Ohio
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - Pennsylvania State Univ / Hershey Med Ctr, Hershey, Pennsylvania
  - Children's Hosp of Philadelphia, Philadelphia, Pennsylvania
  - Univ of Pennsylvania / HIV Clinic, Philadelphia, Pennsylvania
  - Buckley Braffman Stern Med Associates, Philadelphia, Pennsylvania
  - Oncology and Hematology Association, Philadelphia, Pennsylvania
  - Univ of Pittsburgh Med School, Pittsburgh, Pennsylvania
  - Mem Hosp of Rhode Island, Pawtucket, Rhode Island
  - Med Univ of South Carolina, Charleston, South Carolina
  - Univ of Tennessee, Memphis, Tennessee
  - Vanderbilt Univ, Nashville, Tennessee
  - Central Texas Med Foundation, Austin, Texas
  - Dallas Veterans Administration Med Ctr, Dallas, Texas
  - Park Plaza Hosp, Houston, Texas
  - Houston Veterans Administration Med Ctr, Houston, Texas
  - Univ TX Health Science Ctr, Houston, Texas
  - Univ TX San Antonio Health Science Ctr, San Antonio, Texas
  - Med Ctr of Vermont Hosp, Burlington, Vermont
  - Richmond AIDS Consortium, Richmond, Virginia
  - Univ of Washington, Seattle, Washington
  - Univ of Wisconsin, Madison, Wisconsin
- UPR School of Medicine, San Juan, Puerto Rico

REFERENCES:
- [Background] Freimuth WW, Chuang-Stein CJ, Greenwald CA, Cox SR, Edge-Padbury BA, Carberry PA, Wathen LK. Delavirdine (DLV) + didanosine (ddI) combination therapy has sustained surrogate marker response in advanced HIV-1 population. Conf Retroviruses Opportunistic Infect. 1996 Jan 28-Feb 1;3rd:163